CLINICAL TRIAL: NCT07295379
Title: A Retrospective, Single Centre, Observational Study to Evaluate the Safety and Effectiveness of LIQUIBAND FIX8® When Used for Mesh Fixation During Ventral Incisional Hernia Repair.
Brief Title: LIQUIBAND FIX8® for Ventral Incisional Hernia
Acronym: LBF8-03
Status: Not yet recruiting | Type: Observational
Sponsor: Advanced Medical Solutions Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LBF8-03
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hernia Incisional Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All comers: All comers treated with the study device
  Interventions: Device: LIQUIBAND FIX8

INTERVENTIONS:
Device: LIQUIBAND FIX8 — Study device

SUMMARY:
This study is designed to evaluate the safety and performance of device LiquiBand FIX8 Open hernia mesh fixation device. The use of this device is not experimental, as it is already approved for use in the EU (CE-marked). This is a retrospective post market clinical follow-up study to collect information about the use of the device in a real-world setting for ventral incisional hernia repair. Ventral incisional hernias occur following surgery and the most common method of treatment includes implanting a mesh, which in the case of ventral incisional hernia, the standard of care is intra-peritoneal onlay mesh. This is fixed in place using sutures, tacks or adhesive.

The LiquiBand FIX8 Open device is an atraumatic device specifically engineered for strong mesh fixation of hernia repair meshes. Hernia repair meshes are woven sheets of flexible synthetic plastic which are placed tension-free over the weakness in the peritoneum abdominal wall, essentially 'plugging' it up. Tension is created in the abdominal wall during repair, but the mesh allows this tension to be spread out. The mesh must be secured to the underlying tissue and this is often done with the use of tacks or sutures, however, the study device instead uses a glue (N-Butyl 2 cyanoacrylate adhesive) to secure the mesh. The FIX8 Open device is designed for the application of this glue to the implanted hernia repair mesh in order to fix the mesh to the underlying tissue. When the glue is applied to the mesh and tissue, it polymerises (forms a chemical bond) due to the moisture on the tissue surface within approximately 10 seconds and allows the mesh to remain in the correct position. The study device can also be used to close topical wounds (the opening that the surgeon makes on the surface to access the hernia).

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age and ≤ 80 years of age.
* Patient had a ventral incisional hernia (this may include both primary and recurrent).
* Patient underwent a ventral incisional repair and LIQUIBAND FIX8® adhesive was used for mesh fixation (including those patients where supplemental fixation was used)
* Has a minimum of 12 months follow-up.

Exclusion Criteria:

* Every patient who required a ventral incisional hernia repair without concomitant parastomal hernia repair that meets the eligibility criteria will be included in this study. There will be no exclusions specific to the device. Any exclusions relating to device labelling, will have been established as part of the patient's standard of care, prior to the surgical procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All comers for ventral incisional hernia repair at Royal Lancaster Infirmary performed by study Investigator
Sampling Method: Non-Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Performance of LIQUIBAND FIX8 | From surgery to end of follow-up at 12 months
  The performance of LIQUIBAND FIX8® adhesive when used as a method of mesh fixation (independently or in conjunction with another mesh fixation device) during ventral incisional hernia, through reported hernia recurrence rates at 12 months post-surgery.

SECONDARY OUTCOMES:
Reoperation incidence | From surgery to end of follow-up at 12-months
  To evaluate the incidence of reoperation following ventral incisional hernia repair using LIQUIBAND FIX8 as the method of mesh fixation (independently or in conjunction with another mesh fixation device) at discharge, 6-12 weeks follow up and 12 months post-surgery.
SSI incidence | From surgery to end of follow-up at 12-months
  To evaluate the incidence of surgical site infection following ventral incisional hernia repair using LIQUIBAND FIX8 as the method of mesh fixation (independently or in conjunction with another mesh fixation device) at discharge, 6-12 weeks follow up and 12 months post-surgery.
Chronic pain incidence | From surgery to end of follow-up at 12-months
  To evaluate the incidence of chronic pain following ventral incisional hernia repair i.e. beyond 3 months surgery
Adverse Events | From surgery to end of follow-up at 12-months
  To assess post market safety through the reporting of adverse events following ventral incisional hernia repair using LIQUIBAND FIX8 as the method of mesh fixation (independently or in conjunction with another mesh fixation device) at discharge, 6-12 weeks follow up and 12 months post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Lancaster Infirmary, Lancaster, United Kingdom

IPD SHARING:
Plan to Share IPD: No